CLINICAL TRIAL: NCT03394872
Title: Impact of Draining Significant Effusion on Gas Exchange and Lung Mechanics in Patient Under Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Begum Ergan, Staff pulmonologist and intensivist in Department Pulmonary and Critical Care Medicine in Dokuz Eylul Universty Hospital, Dokuz Eylul University, Dokuz Eylul University
Other Study IDs: 2496-GOA
Record Dates: First submitted 2017-12-19; First posted 2018-01-09 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Respiration, Artificial; Pleural Effusion; Ultrasonography
Keywords: Pleural effusion; Mechanical Ventilation; Ultrasonography; Drainage
MeSH Terms: conditions — Respiratory Aspiration; Pleural Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Drainage group: Patients under mechanical ventilator support due to acute respiratory failure who had significant pleural effusion and drainage plan according to the intensive Care Unit (ICU) protocols decided by primary physician
  Interventions: Procedure: Drainage of the pleural effusion

INTERVENTIONS:
Procedure: Drainage of the pleural effusion
  Other Names: Thoracic Ultrasonography performed by USG certificated intensivist to the all subjects included in the study before drainage

SUMMARY:
Patients with acute respiratory failure (ARF) who were receiving mechanical ventilator support, had significant pleural effusion (both transudates and exudates) and drainage plan were evaluated. Decision to drain, timing and duration of drainage were made by primary physician according to the intensive care unit (ICU) protocols.The estimated amount of effusion (mL) was calculated as the maximum pleura-lung distance (mm) x 20 and significant effusion is accepted as ≥ 800 mL according to thoracic ultrasonography (USG) performed by the intensivist. The amount of effusion drained, mechanical ventilator parameters, arterial blood gas results and hemodynamic data were recorded before, at the 1st hour and at the end of drainage up to 30 days after drainage.

ELIGIBILITY:
Inclusion Criteria:

* Patients on mechanical ventilation due to acute respiratory failure
* Estimated effusion > 800 ml according to USG
* Have drainage plan according to ICU protocols decided by primary physician

Exclusion Criteria:

* Have absolute drainage indication (empyema, hemothorax or chylothorax)
* predicted duration of mechanical ventilation less than 72 hours
* contraindications to drainage,
* underlying disease, which prevents lung expansion (chest deformity, central atelectasis)
* malignant effusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critical care patients on mechanical ventilation due to acute respiratory failure and have significant pleural effusion who had drainage plan according to İCU protocols decided by primary physician were enrolled for the study
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Correlation between estimated and drained effusion volume | 1- Estimated effusion volume just before the drainage (by ultrasonography calculated as described in brief summary) 2- Drained effusion volume just after the drainage is terminated up to 30 days after procedure.
  Volume of the effusion estimated and drained was recorded (mL)
Change in Lung mechanics | 1- Dynamic Compliance just before the drainage 2- Dynamic Compliance just after the drainage is terminated up to 30 days after procedure
  Dynamic Compliance (mL/cmH2O)
Change in Oxygenation | 1- PaO2/FiO2 just before the drainage 2- PaO2/FiO2 just after the drainage is terminated up to 30 days after procedure
  PaO2/FiO2 (fraction of inspired oxygen)

CONTACTS AND LOCATIONS:
Overall Officials: Barış Yılmaz, MD, Study Chair — Fellow of Critical Care in Department of Pulmonary and Critical Care Medicine in Dokuz Eylül University; Tuğçe Yılmaz, MD, Study Chair — Fellow of Critical Care in Department of Neurology and Critical Care Medicine in Dokuz Eylül University; Begum Ergan, MD, Principal Investigator — Staff in Department of Pulmonary and Critical Care Medicine in Dokuz Eylül University; Necati Gokmen, MD, Study Director — Staff in Department of Anesthesiology and Critical Care Medicine in Dokuz Eylül University; Kutlay Aydin, MD, Study Chair — Fellow of Critical Care in Department of Anesthsiology and Critical Care Medicine in Dokuz Eylül University

IPD SHARING:
Plan to Share IPD: No